CLINICAL TRIAL: NCT04595188
Title: The Sulphur Amino Acid Requirements in Healthy Adults Over 60 Years
Brief Title: Sulphur Amino Acid Requirements in Adults >60 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Glenda Courtney-Martin, Academic & Clinical Specialist, Project Investigator, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1000071600
Record Dates: First submitted 2020-10-06; First posted 2020-10-20 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Healthy
Keywords: elderly; amino acid requirement; methionine; cysteine; dietary requirement; sulphur amino acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sulphur amino acids in Adults > 60 (Experimental): Total sulphur amino acid, as methionine only: all subjects will receive up to 7 methionine test levels, without dietary cysteine, assigned in random order.
  Minimum methionine, with excess dietary cysteine: all subjects will receive up to 7 methionine test levels, in the presence of excess and constant dietary cysteine, assigned in random order.
  Interventions: Other: Sulphur amino acids

INTERVENTIONS:
Other: Sulphur amino acids — For the total sulphur amino acid requirement, there are 7 different methionine test levels (without dietary cysteine) ranging from 5 to 40 mg of methionine per kilogram body weight per day.
  For the minimum methionine requirement, there are 7 different methionine test levels (with excess dietary cysteine).

SUMMARY:
This study aims to determine the requirements for the sulphur amino acids in adults over the age of 60 years:

1. the total sulphur amino acid requirement as methionine only. Methionine is an essential amino acid.
2. the minimum methionine requirement as methionine in the presence of excess dietary cysteine.

It is known that protein and amino acid metabolism may be altered with age and methionine and cysteine, in particular, may be important in the diet of older adults.

Up to 7 different levels of methionine intake as methionine only (no dietary cysteine) and up to 7 different levels of methionine intake in the presence of excess dietary cysteine will be tested in each subject in random order. Each level of intake will involve a 3-day maintenance diet, with measures being collected on the third.

DETAILED DESCRIPTION:
The sulphur amino acids (SAA) are methionine and cysteine. Methionine is essential and must be obtained from the diet whereas cysteine is considered non-essential and is synthesized from methionine. They have many other important roles that are secondary to their role in protein building. For example, they are needed to make the antioxidant glutathione (GSH), which protects the body's cells from damage. However, protein and GSH metabolism have been shown to change with age and hence, the SAA requirements may also be changed. Despite this, current SAA requirements are based on studies conducted in young adults. Thus, there is a need to determine the SAA requirements directly in older adults.

The purpose of the study is to apply the minimally invasive indicator amino acid oxidation (IAAO) protocol to determine the SAA requirements in healthy adults over 60 years of age. The requirements will be determined as (1) the total sulphur amino acid requirement as methionine only and (2) the minimum methionine requirement by providing methionine in the presence of excess dietary cysteine.

A pre-study assessment will be conducted to assess health status using: medical history and a physical exam; and a blood draw (10mL) for fasting blood glucose and hemoglobin A1c to test for diabetes, vitamin B and folate concentrations, and urea and creatinine to test renal function.

In order to determine the requirements, each participant will be studied at up to 7 varying intakes levels of methionine in random order. Each intake level will be studied over 3-days: two adaptation days (day 1 and 2) and one study day (day 3). On the adaptation days, participants will be provided with a milkshake diet providing all the protein and nutrients they need. Participants will consume 4 meals/day in their usual home environment. On the 3rd day participants will come to the Clinical Research Centre at SickKids where they will be given hourly meals and breath and urine samples at specified times.A blood sample will also be collected for analysis of serum insulin, glucose and secondary parameters (i.e. concentrations of amino acids, glutathione, homocysteine and CRP). The mean (estimate average requirement) total sulphur amino acid requirement and minimum methionine requirement will be calculated with breakpoint analysis using a two-phase linear regression crossover analysis.

ELIGIBILITY:
Inclusion Criteria:

* Consent provided
* Aged 60 to 90 years old
* In good general health as evidenced by medical history, physical health and blood draw
* Fasting blood glucose, hemoglobin A1c (HbA1c), urea, creatinine, vitamin-B6, vitamin- B12 and folate levels within normal ranges for age.
* Willingness to participate in the study.
* BMI <30 kg/m2.

Exclusion Criteria:

* Presence of chronic disease and/or acute illness known to affect protein/amino acid metabolism (e.g. HIV, diabetes, cancer, liver or kidney disease, acute cold or flu)
* Taking medications known to affect protein/AA metabolism (e.g. steroids)
* Inability to tolerate the diet (i.e. allergy)
* Significant weight loss during the past month or consumption of weight reducing diets.
* Significant caffeine consumption (>2 cups per day)
* Significant consumption of alcohol (>1 drink per day i.e. 1 beer or ½ glass of wine).
* Unwilling to have blood drawn from a venous access, or using a ventilated hood indirect calorimeter for the purposes of the study.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Determination of total sulphur amino acid requirements in adults >60 years of age | up to 24 months
  methionine requirement the presence of zero cysteine

SECONDARY OUTCOMES:
Determination of minimum sulphur amino acid requirements in adults >60 years of age | up to 24 months
  methionine requirement in the presence of excess cysteine

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Courtney-Martin, MSc, PhD, RD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paoletti A, Pencharz PB, Ball RO, Kong D, Xu L, Elango R, Courtney-Martin G. The dietary requirement for total sulfur amino acids in adults aged >/=60 years appears to be higher in males than in females. Am J Clin Nutr. 2023 Sep;118(3):538-548. doi: 10.1016/j.ajcnut.2023.06.015. Epub 2023 Jun 24. PMID 37356549